CLINICAL TRIAL: NCT07362849
Title: Construction and Application of the Whole Course Management Scheme for Knee Arthroscopic Ligament Surgery Patients Based on "Internet +"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: KY-2025-154
Record Dates: First submitted 2025-12-11; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Patients Undergoing Knee Arthroscopic Ligament Surgery
Keywords: Construction and application of "Internet plus" full course management model in patients undergoing knee arthroscopic ligament surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group patients were treated and managed using conventional diagnosis and treatment metho (Experimental): On the basis of the conventional diagnosis and treatment mode, the experimental group added an application program for closed-loop management of the entire course of the disease. Within 24 hours of admission, orthopedic specialist nurses conducted personal evaluations of patients, mainly observing their level of importance for postoperative functional exercise, compliance with patients and their families, intention towards the application program, setting personalized goals, providing health guidance, and improving patients' awareness of rehabilitation needs. Teach patients to proficiently use the program's educational video viewing function, function exercise video classification query, upload function exercise videos, view medical feedback, and pay attention to questionnaire filling for in-hospital and post hospital health management. During home stay, orthopedic specialist nurses and rehabilitation therapists conduct weekly assessments of exercise compliance and functional status i
  Interventions: Behavioral: Added applications for closed-loop management of the entire disease course
- Control Group (No Intervention): The control group patients were treated and managed using conventional diagnosis and treatment methods, followed up by telephone calls and follow-up questionnaire surveys for intervention. Routine discharge guidance includes medication guidance, exercise guidance, dietary guidance, and psychological guidance. It guides patients on the precautions, intervention measures, and follow-up time for self-management at home after discharge. Patients are followed up once a month by phone or in person, and questionnaire data is collected during follow-up visits.

INTERVENTIONS:
Behavioral: Added applications for closed-loop management of the entire disease course — Teach patients to proficiently use the program's educational video viewing function, function exercise video classification query, upload function exercise videos, view medical feedback, and pay attention to questionnaire filling for in-hospital and post hospital health management.
  Arms: The control group patients were treated and managed using conventional diagnosis and treatment metho

SUMMARY:
On the basis of the conventional diagnosis and treatment mode, the experimental group added an application program for closed-loop management of the entire course of the disease. Within 24 hours of admission, orthopedic specialist nurses conducted personal evaluations of patients, mainly observing their level of importance for postoperative functional exercise, compliance with patients and their families, intention towards the application program, setting personalized goals, providing health guidance, and improving patients' awareness of rehabilitation needs. Teach patients to proficiently use the program's educational video viewing function, function exercise video classification query, upload function exercise videos, view medical feedback, and pay attention to questionnaire filling for in-hospital and post hospital health management. During home stay, orthopedic specialist nurses and rehabilitation therapists conduct weekly assessments of exercise compliance and functional status in patient uploaded videos. Motivational measures are taken for patients with high cooperation to promote goal achievement. Patients with negative and fatigue attitudes seek professional psychological counseling and provide successful rehabilitation cases to enhance patient confidence. Patients who have doubts during the rehabilitation period outside the hospital can apply the "online information sending mode, online consultation+offline service" in the program. Nurses can help patients register and authenticate, teach them how to use "Zhe Li Nursing Home Service" and place orders online. Orthopedic specialist nurses or rehabilitation therapists can contact the supervising doctor to communicate the patient's needs and provide relevant nursing and rehabilitation technical services on-site. The management backend has functions such as full process traceability of service behavior, workload analysis, and nurse service evaluation. It regularly updates disease-related knowledge within the program, perioperative health education, postoperative functional exercise and intervention measures, and regular functional exercise time reminders. Multi terminal collaboration implements information system integration, establishes a complete electronic health record, and forms a closed-loop management mode throughout the process.

ELIGIBILITY:
Inclusion Criteria:

Orthopedic knee arthroscopic ligament surgery patients; Age range: 18-60 years old; Informed consent from participants in this study; Internet is available at home, and patients and their families can skillfully use mobile WeChat and other functions.

Exclusion Criteria:

Those who give up halfway or have difficulty cooperating to complete the exercise; I am currently participating in other clinical trials that may have an impact on this study; Having a clear history of mental illness and epilepsy in the past; Postoperative complications such as fractures and rheumatoid arthritis (such as thrombosis or osteomyelitis) are present; Lower extremity deep vein thrombosis;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Report on the measurement of knee flexion range of motion (ROM) values for patients treated with knee arthroscopy | 12 weeks
  Use a medical protractor to measure, instruct the patient to lie flat and actively/passively flex to the maximum angle of the knee joint, align the medical protractor with the lateral femoral condyle of the knee joint, align the fixed arm with the longitudinal axis of the femur, and move the measuring arm with the longitudinal axis of the tibia. Record the measurement angle, active range of motion AROM, and passive range of motion PROM

SECONDARY OUTCOMES:
Evaluate daily functional status using Lysholm score after knee arthroscopy treatment | 12 weeks
  The Lysholm score is used for evaluation, which consists of 8 questions with scores ranging from 0 to 100. The higher the score, the better the patient's functional status and their tendency towards daily life activities.

OTHER OUTCOMES:
Evaluate the high and low levels of relevant participants based on the rehabilitation function exercise compliance scale | 12weeks
  The compliance of rehabilitation functional exercise was assessed using the Orthopedic Patient Functional Exercise Compliance Scale developed by Tan Yuanyuan et al. The total score of this scale is 75 points, with ≤ 20 points indicating low compliance, 21-54 points indicating partial compliance, and ≥ 55 points indicating high compliance. The Cronbach's alpha coefficient of the scale is 0.930, and the content validity index is 0.936, which can be used to evaluate the compliance of orthopedic patients with rehabilitation functional exercise.
Evaluate the quality of life level of relevant participants based on the quality of life questionnaire scale | 12weeks
  This study adopts its Chinese version, which includes 5 functional domains, 1 overall quality of life domain, and 9 symptom domains. A higher score in the first two areas indicates a better quality of life, while a higher score in the last area indicates a poorer quality of life. This scale is widely used and has good reliability and validity.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Briggs KK, Lysholm J, Tegner Y, Rodkey WG, Kocher MS, Steadman JR. The reliability, validity, and responsiveness of the Lysholm score and Tegner activity scale for anterior cruciate ligament injuries of the knee: 25 years later. Am J Sports Med. 2009 May;37(5):890-7. doi: 10.1177/0363546508330143. Epub 2009 Mar 4. PMID 19261899
- [Background] Li Y, Gu Z, Ning R, Yin H. Study on the effect of internet plus continuous nursing on functional recovery and medication compliance of patients with knee joint replacement. J Orthop Surg Res. 2023 Jun 11;18(1):424. doi: 10.1186/s13018-023-03907-1. PMID 37303038
- [Background] Backer HC, Wu CH, Schulz MRG, Weber-Spickschen TS, Perka C, Hardt S. App-based rehabilitation program after total knee arthroplasty: a randomized controlled trial. Arch Orthop Trauma Surg. 2021 Sep;141(9):1575-1582. doi: 10.1007/s00402-021-03789-0. Epub 2021 Feb 6. PMID 33547927
- [Background] [13]MA Z L, HUANG Y G, GU X P, et al. Expert consensus on anethesia management of enhanced recovery after adult ambulatory surgery[J]. Medical Journal of Peking Union Medical College Hospital, 2019, 10(6): 562-569. Chinese
- [Background] Jones D, Duffy ME, Flanagan J. Randomized clinical trial testing efficacy of a nurse-coached intervention in arthroscopy patients. Nurs Res. 2011 Mar-Apr;60(2):92-9. doi: 10.1097/NNR.0b013e3182002e46. PMID 21358373
- [Background] Bowman EN, Limpisvasti O, Cole BJ, ElAttrache NS. Anterior Cruciate Ligament Reconstruction Graft Preference Most Dependent on Patient Age: A Survey of United States Surgeons. Arthroscopy. 2021 May;37(5):1559-1566. doi: 10.1016/j.arthro.2021.01.042. Epub 2021 Feb 1. PMID 33539983